CLINICAL TRIAL: NCT02919579
Title: A Placebo- and Active-Controlled Study to Evaluate the Effects of a Single-Dose and Repeat-Administration of Intranasal Esketamine on On-Road Driving in Subjects With Major Depressive Disorder (DriveSaFe2)
Brief Title: A Study to Evaluate the Effects of a Single-Dose and Repeat-Administration of Intranasal Esketamine on On-Road Driving in Participants With Major Depressive Disorder
Acronym: DriveSaFe2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR108228; 2016-002424-86 (EudraCT Number); 54135419TRD1019 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-09-01; First posted 2016-09-29 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Esketamine; Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (7):
- Part A: Sequence ABC (Placebo+Alcohol+Esketamine) (Experimental): Participants will receive intranasal placebo on Day 1 and oral placebo on Day 2 [Treatment A] in Period 1, then intranasal placebo on Day 1 and Oral alcohol on Day 2 [Treatment B] in Period 2, followed by intranasal esketamine on Day 1 and oral placebo on Day 2 [Treatment C] in Period 3.
  Interventions: Drug: Placebo (Intranasal); Drug: Esketamine; Other: Alcohol; Drug: Placebo (Oral)
- Part A: Sequence BCA (Placebo+Alcohol+Esketamine) (Experimental): Participants will receive Treatment B in Period 1, then Treatment C in Period 2, followed by Treatment A in Period 3.
  Interventions: Drug: Placebo (Intranasal); Drug: Esketamine; Other: Alcohol; Drug: Placebo (Oral)
- Part A: Sequence CAB (Placebo+Alcohol+Esketamine) (Experimental): Participants will receive Treatment C in Period 1, then Treatment A in Period 2, followed by Treatment B in Period 3.
  Interventions: Drug: Placebo (Intranasal); Drug: Esketamine; Other: Alcohol; Drug: Placebo (Oral)
- Part A: Sequence CBA (Placebo+Alcohol+Esketamine) (Experimental): Participants will receive Treatment C in Period 1, then Treatment B in Period 2, followed by Treatment A in Period 3.
  Interventions: Drug: Placebo (Intranasal); Drug: Esketamine; Other: Alcohol; Drug: Placebo (Oral)
- Part A: Sequence ACB (Placebo+Alcohol+Esketamine) (Experimental): Participants will receive Treatment A in Period 1, then Treatment C in Period 2, followed by Treatment B in Period 3.
  Interventions: Drug: Placebo (Intranasal); Drug: Esketamine; Other: Alcohol; Drug: Placebo (Oral)
- Part A: Sequence BAC (Placebo+Alcohol+Esketamine) (Experimental): Participants will receive Treatment B in Period 1, then Treatment A in Period 2, followed by Treatment C in Period 3.
  Interventions: Drug: Placebo (Intranasal); Drug: Esketamine; Other: Alcohol; Drug: Placebo (Oral)
- Part B: Placebo+Esketamine (Experimental): Participants will receive intranasal placebo on Day 1, followed by intranasal esketamine on Days 4, 8, 11, 15, 18, 22 and 25.
  Interventions: Drug: Placebo (Intranasal); Drug: Esketamine

INTERVENTIONS:
Drug: Placebo (Intranasal) — Participants will receive intranasal placebo in Part A (as per the treatment sequence in period 1,2 and 3) and Part B.
Drug: Esketamine — Participants will receive intranasal esketamine in Part A (as per the treatment sequence in period 1,2 and 3) and Part B.
Other: Alcohol — Participants will receive oral alcohol in Part A (as per the treatment sequence in period 1,2 and 3).
  Arms: Part A: Sequence ABC (Placebo+Alcohol+Esketamine); Part A: Sequence ACB (Placebo+Alcohol+Esketamine); Part A: Sequence BAC (Placebo+Alcohol+Esketamine); Part A: Sequence BCA (Placebo+Alcohol+Esketamine); Part A: Sequence CAB (Placebo+Alcohol+Esketamine); Part A: Sequence CBA (Placebo+Alcohol+Esketamine)
Drug: Placebo (Oral) — Participants will receive oral placebo in Part A (as per the treatment sequence in period 1,2 and 3).
  Arms: Part A: Sequence ABC (Placebo+Alcohol+Esketamine); Part A: Sequence ACB (Placebo+Alcohol+Esketamine); Part A: Sequence BAC (Placebo+Alcohol+Esketamine); Part A: Sequence BCA (Placebo+Alcohol+Esketamine); Part A: Sequence CAB (Placebo+Alcohol+Esketamine); Part A: Sequence CBA (Placebo+Alcohol+Esketamine)

SUMMARY:
The primary purpose of this study is to evaluate the effect of a single 84-milligram (mg) dose of intranasal esketamine compared to placebo, on next day driving performance and repeated administration of 84 mg intranasal esketamine on same-day driving performance as assessed by the mean difference of standard deviation of lateral position (SDLP) from an on-road driving test.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* If a woman, must have a negative serum beta human chorionic gonadotropin pregnancy test at screening and a negative urine pregnancy test on Day 1 of Period 1 in Part A and prior to study drug administration in Part B
* Comfortable with self-administration of intranasal medication and able to follow instructions provided
* Normal visual acuity (corrected or uncorrected)
* Based on self-report, able to consume an amount of alcohol that typically produces a blood alcohol concentration (BAC) of 0.05 percent (that is, 2 to 3 alcoholic drinks ingested within 2 hours on a single occasion)

Exclusion Criteria:

* Current or prior diagnosis of psychosis/psychotic or bipolar disorder
* Primary sleep disorder, such as insomnia, requiring pharmacological intervention at Screening
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or Day 1 of Period 1 as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12-lead electrocardiogram (ECG) at screening or Day 1 of Period 1 as deemed appropriate by the investigator
* History of moderate or severe use disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV or DSM-5) criteria within 1 year before screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening and Day 1 of Period 1

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
The Effect of a Single 84-Milligram (mg) Dose of Intranasal Esketamine Compared to Placebo, on Next day Driving Performance and Repeated Administration of 84 mg Intranasal Esketamine on Same-day Driving Performance | Part A: Day 2
  Driving performance will be assessed by the mean difference of standard deviation of lateral position (SDLP) from an on-road driving test.
The Effect of a Single 84-mg Dose of Intranasal Esketamine Compared to Placebo, on Next day Driving Performance and Repeated Administration of 84 mg Intranasal Esketamine on Same-day Driving Performance | Part B: Day 1
  Driving performance will be assessed by the mean difference of standard deviation of lateral position (SDLP) from an on-road driving test.
The Effect of a Single 84-mg Dose of Intranasal Esketamine Compared to Placebo, on Next day Driving Performance and Repeated Administration of 84 mg Intranasal Esketamine on Same-day Driving Performance | Part B: Day 11
  Driving performance will be assessed by the mean difference of standard deviation of lateral position (SDLP) from an on-road driving test.
The Effect of a Single 84-mg Dose of Intranasal Esketamine Compared to Placebo, on Next day Driving Performance and Repeated Administration of 84 mg Intranasal Esketamine on Same-day Driving Performance | Part B: Day 18
  Driving performance will be assessed by the mean difference of standard deviation of lateral position (SDLP) from an on-road driving test.
The Effect of a Single 84-mg Dose of Intranasal Esketamine Compared to Placebo, on Next day Driving Performance and Repeated Administration of 84 mg Intranasal Esketamine on Same-day Driving Performance | Part B: Day 25
  Driving performance will be assessed by the mean difference of standard deviation of lateral position (SDLP) from an on-road driving test.

SECONDARY OUTCOMES:
Effect on Subjective Driving Ability Scale | Part A: Day 2; Part B: Day 1, 11, 18 and 25
  Immediately after each driving test, subjects will indicate the perceived quality of their driving performance on a visual analog scale from 0 ('I drove exceptionally poorly') to 20 ('I drove exceptionally well') around a midpoint of 'I drove normally'.
Karolinska Sleepiness Scale (KSS) Score | Part A: Day 2; Part B: Day 1, 11, 18 and 25
  KSS is a participant reported assessment used to rate sleepiness on a scale of 1 to 9, ranging from 'extremely alert' (1) to 'very sleepy, great effort to keep awake, fighting sleep (9).
Efficacy Measured by the Montgomery Asberg Depression Rating Scale (MADRS) | Baseline; Part A: Predose, Day 2; Part B: Predose, Days 1, 11, 18, and 25; End of study (up to Day 98)
  MADRS consists of 10 items covering all the important complaints which Participant with depression have (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Item is scored from 0 (normal) to 6 (severe). Total score (0 to 60) is calculated by adding the scores of all 10 items. A higher score represents a more severe condition. Negative Change in Score Indicates Improvement.
Effects on Suicidal Ideation/Behavior Measured by the Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline; Part A: Predose, Day 2; Part B: Predose, Days 1, 11, 18, and 25; End of study (up to Day 98)
  C-SSRS is a clinician rated assessment of suicidal behavior and / or intent. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 'yes/no' items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Only items with yes responses are listed. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.
Effects on Dissociative Symptoms Using the Clinician-Administered Dissociative State Scale (CADSS) | Baseline; Part A: Predose, Day 1; Part B: Predose, Days 1, 11, 18, and 25
  The CADSS is an instrument for the measurement of present-state dissociative symptoms. The CADSS comprises 23 subjective items, divided into 3 components: Depersonalization, Derealization and Amnesia. Participant's responses are coded on a 5-point scale (0 = "Not at all" through to 4 = "Extremely").
Potential Relationship Between Changes in SDLP and the Plasma Concentration of Esketamine and Noresketamine | Part A: 1 hour postdose (Day 1); Part B: 1 hour postdose (Day 11, 18 and 25)
  Potential relationship will be assessed using visual displays of data. The relationship between the standard deviation of lateral position (SDLP) and the concentration of esketamine and noresketamine in plasma will be evaluated.
Effect on Subjective Mental Effort Scale | Part A: Day 2; Part B: Day 1, 11, 18 and 25
  The level of mental effort the participant had to invest in performing the driving test will be assessed on a 15 centimeter (cm) visual analogue scale with markings ranging from 'absolutely no effort' to over 'extreme effort.
Potential Relationship Between Changes in Mean Lateral Position (MLP) and the Plasma Concentration of Esketamine and Noresketamine | Part A: 1 hour postdose (Day 1); Part B: 1 hour postdose (Day 11, 18 and 25)
  Potential relationship will be assessed using visual displays of data. The relationship between the MLP and the concentration of esketamine and noresketamine in plasma will be evaluated. The MLP will be measured from a validated on-road driving test in a 100 kilometer (km) highway-driving lane.
Potential Relationship Between Changes in Mean Speed and the Plasma Concentration of Esketamine and Noresketamine | Part A: 1 hour postdose (Day 1); Part B: 1 hour postdose (Day 11, 18 and 25)
  Potential relationship will be assessed using visual displays of data. The relationship between the mean speed (MS) and the concentration of esketamine and noresketamine in plasma will be evaluated. The MS will be measured from a validated on-road driving test in a 100 km highway-driving lane.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Leiden, Netherlands

REFERENCES:
- [Derived] Dijkstra FM, van de Loo AJ, Abdulahad S, Bosma ER, Hartog M, Huls H, Kuijper DC, de Vries E, Solanki B, Singh J, Aluisio L, Zannikos P, Stuurman FE, Jacobs GE, Verster JC. The effects of intranasal esketamine on on-road driving performance in patients with major depressive disorder or persistent depressive disorder. J Psychopharmacol. 2022 May;36(5):614-625. doi: 10.1177/02698811221078764. Epub 2022 Feb 25. PMID 35212235
- See also: A Placebo- and Active-Controlled Study to Evaluate the Effects of a Single-Dose and Repeat-Administration of Intranasal Esketamine on On-Road Driving in Subjects With Major Depressive Disorder (DriveSaFe2) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108228&attachmentIdentifier=d2a59202-2675-439e-a1f3-fe2d4c870cd2&fileName=CR108228_CSR_Synopsis.pdf&versionIdentifier=